CLINICAL TRIAL: NCT00203268
Title: An Open Label Pilot Trial to Collect and Evaluate Data on the Use of Dihydroergotamine Mesylate in the Treatment of Two Migraine Attacks Associated With Cutaneous Allodynia
Brief Title: A Study Examining the Use of a Migraine Medicine in the Treatment of Two Migraine Attacks in Patients Who Have Increased Skin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDS/DHE/01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Migraine
Keywords: migraine; cutaneous allodynia
MeSH Terms: conditions — Migraine Disorders | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with dihydroergotamine mesylate (DHE-45) (Experimental): Subjects who treated a moderate to severe migraine 2 and 4 hours after the onset of throbbing headache pain
  Interventions: Drug: dihydroergotamine mesylate

INTERVENTIONS:
Drug: dihydroergotamine mesylate — 1.0 mg. intramuscularly
  Other Names: DHE-45

SUMMARY:
This is a research study examining a migraine medicine dihydroergotamine mesylate (DHE-45).It will be used to treat two migraine attacks in subjects who have a history of skin sensitivity associated with their headaches.This skin sensitivity is called cutaneous allodynia (pronounced q-tay-nee-us al-o-din-ee-uh).Cutaneous allodynia is a sensation of pain when a non-noxious stimulus is applied to normal skin. It has been noted in several studies that in subjects with migraine, seventy nine percent of the subjects experienced allodynia on the facial skin on the same side as the headache. It has also been shown that that once allodynia develops, other migraine medicines that would normally be very effective for migraine pain, become much less effective or ineffective. This study will compare the differences,if any, in attacks treated early with this study drug and treated later with the same study drug. It is hoped that that this trial will provide information on the use of DHE-45 in subjects who have cutaneous allodynia. Understanding more about allodynia may help us understand how the pain system works in migraine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive
* Subjects diagnosed with episodic migraine, with or without aura according to International Headache Criteria (IHS) (Appendix B) for at least one-year prior to screening
* Subjects who experience between 3-10 migraine attacks per month (during the previous 6 months) with no more than 15 days of headache per month.
* Subjects who report their migraine pain quality as pulsating/ throbbing.
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subjects who are able to come for 2-hour in-clinic treatment of two separate migraine attacks
* Subjects who are able to understand and comply with all study procedures.
* Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Pregnant and/or lactating women
* Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects with an abnormal ECG that, in the investigators opinion, would expose them to increased risk of adverse events or interfere with study drug and/or analysis of efficacy/tolerability
* Subjects currently using, or expecting to use during the trial, Cytochrome P450 3A4 (CYP3A4 enzymes) inhibitors (such as protease inhibitors and macrolide antibiotics)
* Subjects with severely impaired hepatic or renal function, as determined by the investigator
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects who currently have or have a history of basilar or hemiplegic migraine
* Subjects who have previously shown hypersensitivity to ergot alkaloids
* Subjects who have a history of non-response to DHE-45, as determined by investigator
* Subjects with uncontrolled hypertension
* Subjects who currently have or who have a history of ischemia and/or vasospastic coronary artery disease
* Subjects who, in the investigators opinion, have significant risk factors of coronary artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Subjects who treated a moderate to severe migraine at 1 hour and at 4 hours after the onset of throbbing pain. Subjects were treated with dihydroergotamine mesylate 1.0 mg. intramuscular (IM). Headache severity was rated by subjects using a 4 point scale : 0=None, 1=mild, 2=moderate, 3=severe
Period: Early Treatment
Arm/Group | Treatment Group
Started | 13
Completed | 9
Not Completed | 4
Not completed — only treated one headache | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: Late Treatment
Arm/Group | Treatment Group
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Subjects who treated a moderate to severe migraine 2 hours and 4 hours after the onset of throbbing pain. Subjects were treated with dihydroergotamine mesylate 1.0 mg. IM. Headache severity was rated by subjects using a 4 point scale : 0=None, 1=mild, 2=moderate, 3=severe.
Arm/Group | Treatment Group
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Headache Relief at the 2 Hour Post Treatment Assessment. Relief Was Measured as a 2-point Change on a 4-point Scale (0=None, 1=Mild, 2=Moderate, 3=Severe)in Both the Early Treatment and Late Treatment Groups.
Description: Data was collected at 2 hours post treatment to assess pain level. This assessment was done when subjects treated a migraine early (defined as treatment at 2 hours after onset of throbbing pain)and then late (defined as treatment at 4 hours after onset of throbbing pain). The proportion of subjects reporting headache relief at the 2 hour post treatment assessment was determined for each group and then compared.
Time Frame: 2 hours post treatment and 4 hours post treatment
Measure: Number; unit: participants
Groups:
- Early Treatment: Subjects who treated a moderate to severe migraine 2 hours after the onset of throbbing pain. Subjects were treated with dihydroergotamine mesylate 1.0 mg. IM. Headache severity was rated by subjects using a 4 point scale : 0=None, 1=mild, 2=moderate, 3=severe.
- Late Treatment: Subjects who treated a moderate to severe migraine 4 hours after the onset of throbbing pain. Subjects were treated with dihydroergotamine mesylate 1.0 mg. IM. Headache severity was rated by subjects using a 4 point scale : 0=None, 1=mild, 2=moderate, 3=severe
Arm/Group | Early Treatment | Late Treatment
Number analyzed (Participants) | 9 | 9
participants
  2 hours post dose | 6 | 5
  4 hours post dose | 6 | 7
Statistical Analysis 1: Comparison: Early Treatment vs Late Treatment; Test type: Superiority or Other; p = .3025, clustered survival analysis

ADVERSE EVENTS:
Arm/Group | Early Treatment | Late Treatment
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/9 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Treatment (N=9) | Late Treatment (N=9)
burning at injection site (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
muscle spasm, quadricep (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Medicinal taste aversion (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No